CLINICAL TRIAL: NCT07158905
Title: A Phase I, Randomized, Double-Blind Study to Evaluate the Safety and Tolerability of AV-1980R in Participants With Preclinical Alzheimer's Disease
Brief Title: AV-1980R (Tau Vaccine) in Preclinical Alzheimer's Disease (TAURUS-1980)
Acronym: TAURUS-1980
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute for Molecular Medicine (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IMM-AV1980R-102; 1R01AG092949-01 (NIH)
Record Dates: First submitted 2025-08-27; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Alzheimer Disease; Preclinical Alzheimer's Disease
Keywords: Tau protein; Immunotherapy; Vaccine; Preclinical Alzheimer's Disease; Alzheimer's Disease; secondary prevention; Neurodegeneration; Preventive Alzheimer's
MeSH Terms: conditions — Alzheimer Disease; Frontotemporal Dementia; Nerve Degeneration

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 3:1 ratio to receive AV-1980R or placebo across three ascending dose cohorts. Each participant gets one assigned intervention in parallel with others.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participants are randomized 3:1 within each cohort to AV-1980R or placebo. Arms reflect three dose levels (20, 60, 180 µg) and a pooled placebo; dosing at Weeks 0, 4, 12, and 36 with follow-up to Week 56.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- AV-1980R 20 µg Arm (Experimental): Participants receive 20 µg AV-1980R intramuscularly at Weeks 0, 4, 12, and 36.
  Interventions: Biological: AV-1980R 20 µg
- AV-1980R 60 µg Arm (Experimental): Participants receive 60 µg AV-1980R intramuscularly at Weeks 0, 4, 12, and 36.
  Interventions: Biological: AV-1980R 60 µg
- AV-1980R 180 µg Arm (Experimental): Participants receive 180 µg AV-1980R intramuscularly at Weeks 0, 4, 12, and 36.
  Interventions: Biological: AV-1980R 180 µg
- Placebo Arm (Placebo Comparator): Participants receive placebo injections (10 mM phosphate buffer with the adjuvant, no antigen) at Weeks 0, 4, 12, and 36.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: AV-1980R 20 µg — MultiTEP-based investigational tau vaccine formulated with the adjuvant. The vaccine is designed to elicit anti-tau antibodies in participants with preclinical Alzheimer's disease.
  Arms: AV-1980R 20 µg Arm
Biological: AV-1980R 60 µg — MultiTEP-based tau vaccine formulated with the adjuvant, 60 µg per dose; intramuscular injections at Weeks 0, 4, 12, and 36; secondary-prevention immunotherapy in preclinical AD.
  Arms: AV-1980R 60 µg Arm
Biological: AV-1980R 180 µg — MultiTEP-based tau vaccine formulated with the adjuvant, 180 µg per dose; intramuscular injections at Weeks 0, 4, 12, and 36; secondary-prevention immunotherapy in preclinical AD.
  Arms: AV-1980R 180 µg Arm
Other: Placebo — 10 mM phosphate buffer formulated with the adjuvant; intramuscular injections at Weeks 0, 4, 12, and 36; no active antigen.
  Arms: Placebo Arm

SUMMARY:
This is a Phase 1, multicenter, randomized, double-blind, placebo-controlled, multiple dose-escalating trial to evaluate the safety, tolerability, and immune response of AV-1980R, an investigational vaccine targeting tau protein, in participants with preclinical Alzheimer's disease. Up to 48 cognitively unimpaired adults aged 65-80 with biomarker evidence of early Alzheimer's disease will be enrolled into three ascending dose cohorts. The study is designed as a secondary prevention trial to test whether therapeutic immunization at the preclinical stage is safe, induces an immune response, and, exploratorily, may favorably affect biomarkers associated with disease progression.

DETAILED DESCRIPTION:
This first-in-human study investigates AV-1980R, a MultiTEP-based active immunotherapy formulated with the adjuvant, as a secondary prevention approach for Alzheimer's disease. The study will randomize up to 48 participants aged 65-80 years in a 3:1 ratio to AV-1980R or placebo across three ascending dose cohorts (20 μg, 60 μg, 180 μg). Participants will receive four intramuscular doses at Weeks 0, 4, 12, and 36, with follow-up through Week 56.

Primary objectives are to evaluate safety and tolerability, monitored by adverse events, labs, ECGs, MRI, and neurological assessments. Secondary objectives include immunogenicity measured by anti-tau antibody titers. Exploratory endpoints include plasma biomarker and tau-PET changes.

ELIGIBILITY:
Inclusion Criteria:

Male or post-menopausal/surgically sterile female, 65-80 years of age.

Cognitively unimpaired with preclinical Alzheimer's disease:

CDR global score = 0. MMSE ≥ 26. WMS-R LM II ≥ 6. Amyloid Probability Score 2 (APS2) > 54 (PrecivityAD2™). Adequate vision/hearing to comply with study procedures. Stable concomitant medications if applicable. Signed informed consent.

Exclusion Criteria:

MRI abnormalities: >1 large lacunar infarct, territorial infarct, >5 microbleeds, ARIA-E, or other significant pathology.

Contraindications to MRI (e.g., pacemaker, metallic implants, severe claustrophobia).

Serious illness or hospitalization within 4 weeks prior to enrollment. Clinically significant cardiovascular, endocrine, hematologic, autoimmune, or neurological disease.

Insulin-dependent diabetes, significant arrhythmias, or seizure disorder. Positive C-SSRS (score ≥ 3). Prior tau or amyloid-beta immunotherapy within 1 year. Immunosuppressive or anticoagulant use that could interfere with study safety. Clinically significant lab abnormalities or positive HIV, HBV, or HCV screening.

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2029-06-15 (Estimated); Study Completion 2029-10-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Baseline through Week 56
  Frequency, severity, and relationship of TEAEs and SAEs; safety assessments include labs, vitals, ECGs, MRI, and neurological exams.

SECONDARY OUTCOMES:
Number of Participants with Clinically Significant Changes in Vital Signs | Baseline through Week 56
  Number of participants with clinically significant abnormalities or changes in blood pressure, heart rate, respiratory rate, or body temperature.
Number of Participants with Clinically Significant Changes in ECG Results | Baseline through Week 56
  Number of participants with new or worsening clinically significant ECG abnormalities.
Number of Participants with Clinically Significant Changes in Laboratory Tests | Baseline through Week 56
  Number of participants with new or worsening abnormalities in hematology, serum chemistry, coagulation, or urinalysis results.
Number of Participants with Clinically Significant Changes in Physical Examinations | Baseline through Week 56
  Number of participants with new or worsening abnormal findings on physical examination.
Number of Participants with Clinically Significant Changes in Neurological Examinations | Baseline through Week 56
  Number of participants with new or worsening abnormal neurological findings.
Incidence of Amyloid-Related Imaging Abnormalities (ARIA-E and ARIA-H) | Baseline through Week 56
  Number of participants with vasogenic edema (ARIA-E), effusions, ischemic events, hemorrhagic events, or associated clinical symptoms detected on MRI.
Change from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline, Weeks 12, 36, 40, and 56
  Change from baseline in suicidality assessment using the Columbia-Suicide Severity Rating Scale (C-SSRS; range: 0-25, with higher scores indicating greater severity of suicidal ideation and behavior).
Change from Baseline in Serum Anti-Tau Antibody Concentrations | Baseline through Week 56
  Quantification of anti-tau antibody titers induced by AV-1980R vaccination.
Detection of T Helper (Th) Cell Responses Specific to MultiTEP Platform | Baseline through Week 56
  Presence of antigen-specific Th cell responses against the MultiTEP vaccine platform.
Detection of Autoreactive Th-Cell Responses Specific to Tau | Baseline through Week 56
  Presence of autoreactive Th cell responses directed against tau epitopes.

OTHER OUTCOMES:
Change from Baseline in Plasma Biomarker Concentrations (pg/mL) | Baseline through Week 56
  Change in plasma concentrations of Aβ42, Aβ40, pTau217, pTau181, pTau231, total tau (t-tau), neurofilament light (NfL), and glial fibrillary acidic protein (GFAP), reported in pg/mL.
Change from Baseline in Immunoglobulin Isotypes and Subclasses (mg/dL) | Baseline through Week 56
  Change in serum concentrations of IgM, total IgG, and IgG subclasses (IgG1, IgG2, IgG3, IgG4), reported in mg/dL
Phenotyping of Activated T Cells | Baseline through Week 56
  Characterization of activated T cell subsets by flow cytometry.
T Cell Proliferative Response | Baseline through Week 56
  Assessment of proliferative capacity of T cells following antigen stimulation.
Polarization of Cellular Responses | Baseline through Week 56
  Cytokine production by activated T cells to evaluate polarization of Th1/Th2/Th17 responses.
Change from Baseline in Plasma Biomarker Ratios | Time Frame: Baseline through Week 56
  Change in plasma biomarker ratios including Aβ42/40 ratio and Aβ42/tau ratios (unitless)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Agadjanyan, PhD, Principal Investigator — Institute MM; Roman Kniazev, Study Director — Institute MM
Locations (1):
- Comprehensive Center for Brain Health, Boca Raton, Florida, United States

IPD SHARING:
Plan to Share IPD: No